CLINICAL TRIAL: NCT00568347
Title: Evaluation of the Effects of Varying Doses of Inhaled Corticosteroids on Suppression of Total Exhaled, Bronchial, and Alveolar Nitric Oxide as Markers of Endogenous Inflammation in Patients With Moderate-to-severe COPD
Brief Title: Evaluation Inhaled Corticosteroids on Exhaled Nitric Oxide Gas Exchange
Status: Completed | Type: Observational
Sponsor: Arthur F Gelb MD (Individual)
Responsible Party: Sponsor-Investigator, Arthur F Gelb MD, Arthur F Gelb MD, Gelb, Arthur F., M.D.
Organization: Gelb, Arthur F., M.D. (Individual)
Other Study IDs: 20061697A; NCT00569348 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: COPD
Keywords: chronic airflow obstruction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- long acting bronchodilator: salmeterol 50mcg bid by DPI, no fluticasone in patients with COPD/emphysema to evaluate effect on bronchodilation and exhaled nitric oxide
  Interventions: Drug: Salmeterol
- bronchodilator/ inhaled corticosteroid: fluticasone 250mcg/salmeterol 50 mcg bid X 3momths to evaluate effect on lung function and exhaled nitric oxide
  Interventions: Drug: fluticasone 250/salmeterol 50; Drug: salmeterol and fluticasone propionate
- C: Fluticasone 100mcg/salmeterol 50mcg
  Interventions: Drug: fluticasone 100mcg/ salmeterol 50mcg; Drug: salmeterol

INTERVENTIONS:
Drug: fluticasone 100mcg/ salmeterol 50mcg — inhaled fluticasone 100mcg/salmeterol 50mcg bid X 3 months
  Other Names: Advair 100/50
  Groups: C
Drug: fluticasone 250/salmeterol 50 — inhaled fluticasone 250/salmeterol 50 X 3 months to evaluate effect on lung function and exhaled nitric oxide
  Other Names: Advair 250/50
  Groups: bronchodilator/ inhaled corticosteroid
Drug: salmeterol — salmeterol 50 mcg by dry powder inhaler disk bid to evaluated effect on lung function and exhaled nitric oxide
  Other Names: Serevent 50mcg
  Groups: C
Drug: Salmeterol — salmeterol 50mcg bid X 3months
  Other Names: serevent 50 mcg disk
  Groups: long acting bronchodilator
Drug: salmeterol and fluticasone propionate — salmeterol 50mcg/fluticasone 250mcg by DPI bid
  Other Names: Advair 250/50
  Groups: bronchodilator/ inhaled corticosteroid

SUMMARY:
To evaluate the role of inhaled corticosteroids to suppress nitric oxide gas exchange in stable patients with moderate-to-severe COPD who are current non-smokers and not on oral corticosteroids.

DETAILED DESCRIPTION:
Stable, non-smoking COPD patients not on oral corticosteroids will be randomized in single blinded study to evaluate nitric oxide gas exchange at baseline, and subsequent effects of fluticasone 100mcg/salmeterol 50mcg bid, and fluticasone 250mcg/salmeterol 50mcg bid. Primary end points will include measurements of nitric oxide at varying expiratory flow rates to calculate bronchial, and small airway/alveolar nitric oxide. Secondary end points will evaluate lung function. Exhaled nitric oxide production presumably reflects endogenous inflammation. Normal healthy, non-smoking controls will be used for comparison, with exhaled nitric oxide measured before and after 3 weeks of low dose inhlaed corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of copd
* Current non-smoker
* Not on oral corticosteroids
* Must be able to use Advair discus or salmeterol discus

Exclusion Criteria:

* Pregnancy
* Current smoker
* On corticosteroids
* Clinically unstable

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
total exhaled, bronchial, and small airway/alveolar nitric oxide | 3 months

SECONDARY OUTCOMES:
lung function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Gelb, MD, Principal Investigator — Arthur F Gelb Medical Corporation
Locations (1):
- Arthur F Gelb MD, Lakewood, California, United States

REFERENCES:
- [Result] Gelb AF, Flynn Taylor C, Shinar C. Nitric Oxide gas exchange in COPD. Am J Respir Crit Care Med 2007; 174: A630.
- [Derived] Gelb AF, George SC, Camacho F, Fraser C, Flynn Taylor C, Shakkottai S. Increased nitric oxide concentrations in the small airway of older normal subjects. Chest. 2011 Feb;139(2):368-375. doi: 10.1378/chest.10-1157. Epub 2010 Aug 12. PMID 20705799
- [Derived] Gelb AF, Flynn Taylor C, Krishnan A, Fraser C, Shinar CM, Schein MJ, Osann K. Central and peripheral airway sites of nitric oxide gas exchange in COPD. Chest. 2010 Mar;137(3):575-84. doi: 10.1378/chest.09-1522. Epub 2009 Oct 9. PMID 19820080